CLINICAL TRIAL: NCT05011188
Title: A Phase 1b/2 Study of FOR46 in Combination With Enzalutamide in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: FOR46 in Combination With Enzalutamide in Patients With Metastatic Castration Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rahul Aggarwal (Other)
Collaborators: Fortis Therapeutics, Inc. (Industry); Kyntra Bio (Industry)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21555; NCI-2021-08857 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Prostate Cancer
Keywords: FOR46; Enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Immunoconjugates; enzalutamide; pegfilgrastim; Granulocyte Colony-Stimulating Factor; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Does Escalation (Experimental): Approximately 3 dose levels of FOR46 will be evaluated. Participants will receive a lead-in treatment period of enzalutamide monotherapy for 14 days (day -14 to day -1), followed by addition of FOR46 on Cycle 1 Day 1. If participants are on enzalutamide at the time of study entry, and remain on continuous dosing at 160 mg daily, the lead-in treatment period will not be required. Prophylactic Pegfilgrastim (G-CSF) 6mg, subcutaneously (SQ) will also be administered on Day 2 during all treatment cycles. Pegfilgrastim could be modified to a lower dose of 3 mg with treating investigator approval.
  Interventions: Biological: FOR46; Biological: Enzalutamide; Drug: Pegfilgrastim; Procedure: Blood Samples
- Dose Expansion (Experimental): Participants will receive a lead-in treatment period of enzalutamide monotherapy for 14 days (day -14 to day -1), followed by addition of FOR46 on Cycle 1 Day 1, at the maximum tolerated dose (MTD) as determined in Phase 1b. If participants are on enzalutamide at the time of study entry, and remain on continuous dosing at 160 mg daily, the lead-in treatment period will not be required. Prophylactic Pegfilgrastim (G-CSF) 6mg, subcutaneously (SQ) will also be administered on Day 2 during all treatment cycles. Pegfilgrastim could be modified to a lower dose of 3 mg with treating investigator approval.
  Interventions: Biological: FOR46; Biological: Enzalutamide; Drug: Pegfilgrastim

INTERVENTIONS:
Biological: FOR46 — Given intravenously (IV)
  Other Names: Antibody-Drug Conjugate (ADC); anti-CD46 antibody conjugate
Biological: Enzalutamide — Given orally (PO)
  Other Names: XTANDI
Drug: Pegfilgrastim — Given subcutaneously (subQ)
  Other Names: G-CSF
Procedure: Blood Samples — Blood samples will be taken for correlative studies
  Other Names: Blood Specimen; Biospecimen
  Arms: Does Escalation

SUMMARY:
This is a Phase 1b/2 study evaluating FOR46 in combination with enzalutamide in patients with metastatic castration resistant prostate cancer (mCRPC) after prior progression on abiraterone. FOR46 is designed to target and bind to CD46, a transmembrane cellular protein expressed at moderate or high levels in numerous cancer types. The investigators hypothesize that the combination of FOR46 plus enzalutamide will achieve a clinically significant composite response rate with sufficient durability of response in mCRPC patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Phase 1b:

I. To determine the maximally tolerated dose (MTD) and recommended phase 2 dose (RP2D) of FOR46 in combination with enzalutamide in patients with mCRPC.

Phase 2:

I. To determine the composite response rate of FOR46 plus enzalutamide, defined as:

1. Decline in serum PSA >= 50% (PSA50) from baseline, confirmed by repeat measurement at least 4 weeks later, and/or
2. Objective response by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.

SECONDARY OBJECTIVES:

Phase 1b and Phase 2:

I. To determine the PSA50 response rate.

II. To determine the objective response rate by RECIST 1.1 criteria among patients with measurable soft tissue by RECIST 1.1 criteria at baseline.

III. To determine the median duration of objective response.

IIII. To determine the median time to prostate-specific antigen (PSA) progression by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria.

V. To determine the median radiographic progression-free survival by PCWG3 criteria.

VI. To determine the median overall survival.

VII. To determine the safety of the combination.

OUTLINE:

Participants may continue study treatment from the time of treatment initiation until confirmed radiographic disease progression per PCWG3 / RECIST 1.1 criteria, unequivocal clinical progression, unacceptable toxicity, or patient withdrawal, whichever occurs first. Patients will be followed for overall survival every 90 days (+/- 30 days) from last dose of study treatment, until death, withdrawal of consent, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic prostate adenocarcinoma.
2. Disease progression by PCWG3 criteria at study entry.
3. Prior progression by PCWG3 criteria on one or more androgen signaling inhibitors including abiraterone acetate, enzalutamide, apalutamide, and/or darolutamide.
4. No prior taxane-based chemotherapy for the treatment of mCRPC. Prior taxane use in the castration-sensitive prostate cancer (CSPC) setting allowed provided last dose > 6 months prior to study entry.
5. Patients must be evaluable for the primary endpoint of composite response, and must have either serum PSA ≥ 2 ng/mL during Screening and/or measurable disease by RECIST 1.1 criteria.
6. Participants must be willing to undergo metastatic tumor biopsy during Screening. If there is no safely accessible metastatic lesion, this requirement will be waived.
7. Dose Expansion only: Participants must be willing to undergo CD46-directed Positron Emission Tomography (PET) imaging during Screening (Co-enrolling on NCT05245006, Groups B and C)
8. Castrate level of serum testosterone at study entry (<50 ng/dL). Patients without prior bilateral orchiectomy are required to remain on Luteinizing hormone-releasing hormone (LHRH) analogue treatment for duration of study.
9. No other systemic anti-cancer therapies administered other than LHRH analogue within 14 days or, 5 half-lives, whichever is shorter, prior to initiation of study treatment. Adverse events related to prior anti-cancer treatment related to therapies other than LHRH analogue must have recovered to Grade ≤ 1 with the exception of any grade alopecia. a. Patients receiving enzalutamide prior to study entry may continue treatment at their current enzalutamide dose level without requirement for wash-out period.
10. Age >=18 years.
11. Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky performance status >= 70 percent (%)).
12. Demonstrates adequate organ function as defined below:

    1. Absolute neutrophil count ≥ 1,500/microliter (mcL).
    2. Platelets >= 100,000/mcL and no platelet transfusions during the 14 days prior to first dose of FOR46.
    3. Hemoglobin >= 8.0 grams per deciliter (g/dL) without red blood cell transfusion during the 14 days prior to first dose of FOR46.
    4. Total bilirubin <=1.5 x institutional upper limit of normal (ULN), unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits.
    5. Aspartate aminotransferase (AST) /serum glutamic-oxaloacetic transaminase (SGOT) <=3 x institutional institutional upper limit of normal (ULN).
    6. Alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) =3 x ULN.
    7. Serum creatinine <= 1.5 x institutional upper limit of normal OR Calculated creatinine clearance glomerular filtration rate (GFR) >= 60 mL/min, calculated using the Cockcroft-Gault equation.
    8. Serum sodium level >=130 mmol/L.
13. Ability to understand a written informed consent document, and the willingness to sign it.
14. Individuals with concurrent second malignancy requiring active treatment at study entry. Nonmelanoma skin cancer, non-muscle invasive bladder cancer, and other carcinomas-in-situ are allowable exceptions.
15. Patients must agree to use adequate contraception prior to the study, for the duration of study participation, and 60 days after last administration of study treatment. Adequate contraception includes:

    1. Patients who are sexually active should consider their female partner to be of childbearing potential if she has experienced menarche and is not postmenopausal (defined as amenorrhea > 24 consecutive months) or has not undergone successful surgical sterilization. Even women who use contraceptive hormones (oral, implanted, or injected), an intrauterine device, or barrier methods (diaphragms, condoms, spermicide) should be considered to be of childbearing potential.
    2. Acceptable methods of contraception include continuous total abstinence, or double-barrier method of birth control (e.g. condoms used with spermicide, or condoms used with oral contraceptives). Periodic abstinence and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Has received prior radiotherapy within 2 weeks of first dose of FOR46.
2. Prior treatment with FOR46 or another CD46-targeting therapeutic agent.
3. Prior histologic evidence of de novo or treatment-emergent small cell neuroendocrine prostate cancer. Pathologic assessment of baseline tumor biopsy performed during Screening is not required for determination of study eligibility.
4. Cardiac condition as defined as one or more of the following:

   1. Uncontrolled supraventricular arrhythmia or ventricular arrhythmia requiring treatment.
   2. New York Heart Association (NYHA) congestive heart failure class III or IV.
   3. History of unstable angina, myocardial infarction, or cerebrovascular accident within 6 months prior to Cycle 1, Day 1.
5. History of seizure or pre-disposing condition including:

   1. History of brain metastasis.
   2. Cerebrovascular accident (CVA) within 6 months prior to study entry.
   3. History of intracranial hemorrhage.
6. History of pneumonitis.
7. Is receiving systemic steroid therapy at a prednisone equivalent dose of > 10 milligram daily or other form of immunosuppressive therapy within 7 days prior to first dose of study drug.
8. Has an active infection requiring intravenous antibiotics within 7 days prior to Cycle 1, Day 1.
9. Use of a prohibited concomitant medication within 7 days of first dose of FOR46, including:

   a. Strong inhibitor of CYP3A4 (boceprevir, clarithromycin, cobicistat, conivaptan, diltiazem, danoprevir/ritonavir, elvitegravir/ritonavir, grapefruit juice, idelalisib, indinavir/ritonavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, paritaprevir/ritonavir/ombitasvir and/or dasabuvir, posaconazole, ritonavir, saquinavir/ritonavir, tipranavir/ritonavir, troleandomycin, and voriconazole).
10. Major surgery within 28 days prior to Cycle 1, Day 1. Minor procedures including biopsies, dental surgery, cataract surgery, or outpatient procedure are allowed.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) (Phase 1b) | Up to 3 weeks
  A minimum of 3 patients will be treated at each dose level. If < 33%of patients (i.e. 0 of 3 patients, or 1 of 6 patients) within a cohort have a dose-limiting toxicity (DLT in Cycle 1, then enrollment of the next cohort may commence upon approval of Data and Safety Monitoring Committee. At any dose level, dose escalation will be discontinued if >= 2 of 3 to 6 patients within a cohort experience a DLT in Cycle 1, the MTD will have been exceeded. The previous dose level will then be considered the MTD if 6 patients were previously evaluated at this dose level. If this dose level was previously evaluated with 3 patients, then 3 additional patients will be enrolled at this dose level; if 0 or 1 of the additional 3 patients experiences a DLT in Cycle 1, then this dose level will be considered the MTD.
Number of participants with Dose-Limiting Toxicities (Phase 1b) | Up to 3 weeks
  Dose-limiting toxicities classified using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0will be tabulated by dose level and reported in descriptive fashion.
Composite response rate (CRR) (Phase 2) | Up to 2 years
  Composite response is defined as a >= 50% decline from baseline PSA (defined by Cycle 1 Day 1 value), confirmed by repeat measurement >= 4 weeks later AND/OR objective tumor response by RECIST 1.1 criteria The composite response rate along with 95% confidence interval will be reported

SECONDARY OUTCOMES:
Proportion of participants with a greater than or equal to 50% change in PSA (PSA50) | Up to 2 years
  PSA50 response is defined as above, a ≥ 50% decline from baseline in serum PSA, confirmed by repeat measurement ≥ 4 weeks later. The PSA50 response proportion will be reported along with 95% confidence interval for each study cohort, for the subset of PSA-evaluable patients (serum PSA ≥ 2 ng/mL at baseline)
Objective response rate (ORR) | Up to 2 years
  The objective response rate and median duration of response will be reported along with 95% confidence interval for the subset of patients with measurable soft tissue disease by RECIST 1.1 criteria at baseline
Median duration of objective response | Up to 2 years
  The median duration of response will be reported along with 95% confidence interval for the subset of patients with measurable soft tissue disease by RECIST 1.1 criteria at baseline
Median time to PSA progression | Up to 2 years
  Median time to PSA progression assessed by PCWG3 criteria will be determined from the date of first dose of protocol-defined therapy, using Kaplan-Meier product limit method. Patients who discontinue treatment for reasons other than adverse event, patient withdrawal, etc. will be censored by the date of last treatment.
Median radiographic progression-free survival | Up to 2 years
  Median radiographic progression-free survival assessed by PCWG3 criteria will be determined from the date of first dose of protocol-defined therapy, using Kaplan-Meier product limit method. Patients who discontinue treatment for reasons other than adverse event, patient withdrawal, etc. will be censored by the date of last treatment.
Median overall survival survival. | Up to 2 years
  The median overall survival along with 95% confidence interval will be determined from the date of first dose of protocol-defined therapy until death from any cause, using the Kaplan-Meier product limit method. Patients will be followed for long-term survival as outlined in the Study Procedures. Patients who withdraw from study will be censored for analysis of overall survival using the date of study withdrawal.
Frequency of treatment-related, adverse events (AE) | Up to 2 years
  Adverse events will be recorded and severity graded using CTCAE version 5.0. The frequency and highest grade of severity of adverse events will be descriptively reported

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No